CLINICAL TRIAL: NCT06394843
Title: Mobilization of Fluid and Fluid Currents During Hemodialysis
Brief Title: Fluid Currents During Hemodialysis
Status: Not yet recruiting | Type: Observational
Sponsor: Joachim Zdolsek (Other)
Collaborators: Region Östergötland (Other)
Responsible Party: Sponsor-Investigator, Joachim Zdolsek, Associate professor, Principal investigator, University Hospital, Linkoeping
Organization: University Hospital, Linkoeping (Other)
Other Study IDs: MVVH
Record Dates: First submitted 2024-04-15; First posted 2024-05-01 (Actual); Last update posted 2024-05-01 (Actual); Status verified 2024-04

CONDITIONS: Patients Undergoing Hemodialysis
Keywords: Hemodialysis
MeSH Terms: interventions — Ultrafiltration

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- <500 ml Ultrafiltration: Patients undergoing hemodialysis with less than 500 ml ultrafiltration
  Interventions: Other: Ultrafiltration
- >2000 ml Ultrafiltration: Patients undergoing hemodialysis with than 2000 ml ultrafiltration
  Interventions: Other: Ultrafiltration

INTERVENTIONS:
Other: Ultrafiltration — Patients are selected depending on need of ultrafiltration

SUMMARY:
During dialysis, three objectives are achieved. 1. Blood is cleansed from waste products. 2. Excess water is removed. 3. Electrolytes are regulated. These processes occur simultaneously but vary from patient to patient depending on their specific needs. Some patients still produce urine, but of poor quality. Others have no residual urine production at all and require removal of fluid from both blood and tissues. Hypotension may occur during dialysis, related to intravascular hypovolemia and inadequate fluid reinfusion, which is common during ultrafiltration exceeding 400 ml/h. The amount of fluid removed is influenced by fluid recruitment from tissues. This mainly occurs in two different ways: osmotic recruitment across capillary membranes from the perivascular space or via lymphatic reflow. The proportions are not fully understood. When fluid is recruited from the perivascular space, the influx of albumin and immunoglobulins is unlikely. However, these should accompany lymph to the blood if lymphatic flow is increased. The content of albumin and immunoglobulins differs between lymph and plasma. Thus, the proportions of fluid recruitment from tissues should be calculable using mass balance calculations based on ultrafiltrate, colloid osmotic pressure, hemoglobin, albumin, and immunoglobulin concentrations. The rate and proportions of fluid reinfusion into the bloodstream are not fully understood. Therefore, in this study, the aim is to monitor fluid reinfusion and its proportions of lymph/osmotic recruitment into the bloodstream.

DETAILED DESCRIPTION:
In Sweden, approximately 3200 patients undergo hemodialysis annually. In some cases, it is solely about blood purification, but for many patients, removal of excess fluid accumulated since the last dialysis treatment is also necessary. The amount of fluid removal/ultrafiltration prescribed by the physician during dialysis primarily depends on the amount of residual urine the patient produces but also on the patient's fluid intake between dialysis treatments. The most common complication of hemodialysis is hypotension during treatment, occurring in about 10% of treatment sessions according to previous studies. These hypotensive episodes lead to temporary hypoperfusion, and repeated episodes can cause permanent organ damage. The main cause of these hypotensive episodes is the reduction in circulating volume during ultrafiltration, i.e., fluid removal. The excess fluid that the patient accumulates between treatments is mainly located outside the bloodstream. Therefore, in connection with fluid removal during hemodialysis, there is compensatory fluid recruitment to the circulation, increasing the circulating volume and preventing hypotension. How this occurs and from which fluid compartment fluid is recruited is not yet mapped out. To increase understanding of hemodialysis and optimize treatment while minimizing the risk of hypotension, it is interesting to understand how fluid recruitment occurs and from which fluid compartments recruitment occurs. Using fluid kinetic calculations, it has been possible to measure whether fluid is recruited perivascularly or from the lymphatic system during albumin infusion depending on the concentrations of proteins such as IgG and IgM, as their concentrations differ. By measuring the concentrations of these proteins in blood samples over time, it has been possible to calculate from which fluid compartment fluid has been recruited.

Purpose and Objective

The aim is to study:

* How much fluid is drawn from the interstitial space during dialysis, depending on whether fluid removal is needed or not.
* The size and rate of fluid reinfusion during ongoing dialysis.
* The composition of the recruited fluid from the interstitium, i.e., the proportion consisting of lymph/lymph reflow and the proportion recruited across capillary membranes/venulae from the pericapillary space.

Hypotheses The null hypothesis is that no detectable difference in fluid flows or source of fluid recruitment is found, between patients where a large volume is dialyzed and those patients who do not have significant fluid removal during dialysis.

The alternative hypothesis is that a clinical relevant difference in fluid flows from the interstitium and the pathway for fluid recruitment to the bloodstream is detected.

Outcome Measures

Primary outcome variables are:

Recruitment of fluid from the interstitium calculated from fluid removal and hemoglobin changes. Proportion of recruited fluid via lymph or via capillary/venulae walls based on fluid recruitment and changes in plasma albumin and immunoglobulins G and M.

Secondary outcome variables are:

Weight, blood pressure impact, and changes in bioimpedance variables.

Study Design:

Open-label, prospective clinical observational study, where patients are divided into two groups. One group with an intact urine production, and dialysis is performed solely to "cleanse" the blood and second group with little or no urine production, which requires significant fluid removal, in addition to blood purification, .

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing hemodialysis (<500 ml or >2000 ml ultrafiltration)

Exclusion Criteria:

* Patients who may be affected by blood sampling, i.e., have low hemoglobin concentration independent of dilution before dialysis (Hb 85 g/L).
* Patients who drink large amounts of water during regular dialysis (> 2 glasses, approximately 0.5 L).

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing hemodialysis regularly at the dialysis department at Vrinnevisjukhuset in Norrköping are screened if they are expected to meet the inclusion criteria for the study. Those who meet the inclusion criteria and have no exclusion criteria are asked to participate.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2024-05-06 (Estimated); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Proportion of fluid recruited via endothelial wall vs lymph | 8 hours
  Recruitment of fluid from the interstitium calculated from fluid removal and hemoglobin changes. Proportion of recruited fluid via lymph or via capillary/venulae walls based on fluid recruitment and changes in plasma albumin and immunoglobulins G and M

SECONDARY OUTCOMES:
Weight | 8 hours
  Weight (before and after hemodialysis)
Blood pressure | 8 hours
  Impact of hypovolemia related to ultrafiltration on blood pressure
Bioimpedance | 8 hours
  Change in Bioimpedance related to hemodialysis

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan Bodare, MD, Principal Investigator — Region Oestergoetland; Erik Golsäter, MD, Principal Investigator — Region Oestergoetland; Fredrik Sundelin, MD, Principal Investigator — Region Oestergoetland
Locations (1):
- Vrinnevi Hospital, Norrköping, Östergötland County, Sweden

IPD SHARING:
Plan to Share IPD: Yes
Results will be presented in an international medical journal
Supporting Information: CSR
Time Frame: Approximately 6 to 12 months after completion of the study.

REFERENCES:
- [Background] Zdolsek JH, Zdolsek M, Hahn RG. Recruitment of efferent lymph during infusion of 20 % albumin. Microvasc Res. 2023 Jul;148:104539. doi: 10.1016/j.mvr.2023.104539. Epub 2023 May 6. PMID 37156370

DOCUMENTS (2):
  • Study Protocol (2024-03-21): https://cdn.clinicaltrials.gov/large-docs/43/NCT06394843/Prot_000.pdf
  • Statistical Analysis Plan (2024-03-21): https://cdn.clinicaltrials.gov/large-docs/43/NCT06394843/SAP_001.pdf